CLINICAL TRIAL: NCT00473161
Title: Use of Surface Electromyography Biofeedback to Improve Reaching in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Other Study IDs: EMG biofeedback
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Cerebral Palsy; Weakness; Hypertonia
Keywords: movement disorders; childhood
MeSH Terms: conditions — Cerebral Palsy; Asthenia; Muscle Hypertonia; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: surface EMG biofeedback

SUMMARY:
A newly-developed device for biofeedback of surface EMG will be used to either increase or decrease activity in the muscles of children with poor reaching due to cerebral palsy.

DETAILED DESCRIPTION:
Children ages newborn to 21 with a diagnosis of arm weakness, hypertonia, or hyperkinesia due to cerebral palsy will be recruited. A muscle that is either over-active or under-active will be selected for each child. The child will be provided with the device to wear for 1 month in order to call attention to the identified muscle. At the beginning and end of the month, reaching will be assessed using three-dimensional kinematic motion capture. The outcome measure will be the speed and curvature of reaching to a target in front of the child.

ELIGIBILITY:
Inclusion Criteria:

* weakness, hypertonia, or hyperkinetic disorder affecting one or both arms
* reduced speed or quality of reaching

Exclusion Criteria:

* any condition that would increase the risk of participation

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with movement disorders, cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence D Sanger, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States